CLINICAL TRIAL: NCT06102928
Title: A Prospective, Multicenter, Single-arm Clinical Study of the Combination of Anlotinib and Aumolertinib in the First-line Treatment of Advanced Non-small Cell Lung Cancer With EGFR 21L858R Mutation
Brief Title: A Clinical Study of the Combination of Anlotinib and Aumolertinib in the First-line Treatment of Advanced NSCLC With EGFR 21L858R Mutation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yuqi Cheng, Professor Jianqing zhang, Kunming Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC202316
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Non-Small Cell Lung Cancer With Mutation in Epidermal Growth Factor Receptor
Keywords: non-small cell lung cancer;anlotinib;aumolertinib;combined therapy;efficacy
MeSH Terms: interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Participants who met the study protocol were treated with anlotinib and aumolertinib.Aumolertinib mesylate tablets are administered 110 mg orally once a day until disease progression or unacceptable toxicity. Anlotinib hydrochloride capsules were given 12 mg once a day, taken for 2 weeks and then discontinued for 1 week, with a treatment cycle every 21 days. If grade 3 or above treatment-related toxicity occurs, anlotinib can be reduced to 10 mg or 8 mg once daily until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Combined therapy of anlotinib and aumolertinib

INTERVENTIONS:
Drug: Combined therapy of anlotinib and aumolertinib — Participants were treated with anlotinib and aumolertinib.Aumolertinib mesylate tablets are administered 110 mg orally once a day,and anlotinib hydrochloride capsules were given 12 mg once a day, taken for 2 weeks and then discontinued for 1 week, with a treatment cycle every 21 days. If grade 3 or above treatment-related toxicity occurs, anlotinib can be reduced to 10 mg or 8 mg once daily.

SUMMARY:
This study is a prospective, multicenter, single arm clinical study. Thirty subjects who will have been diagnosed with locally advanced or metastatic non-small cell lung cancer with EGFR 21L858R mutation detected in lung cancer tissue or peripheral blood will be recruited and treated with anlotinib and aumolertinib. The efficacy will be evaluated according to the Solid Tumor Efficacy Evaluation Standard (RECIST 1.1), and evaluated every 6 to 8 weeks. The survival status and adverse reactions of the subjects will be recorded. The study will be terminated when the subjects experience disease progression or intolerable drug toxicity, or the subjects withdraw their informed consent. The main purpose of the study is to observe the efficacy and safety of the combined treatment regimen in such subjects. The primary endpoint of the study is median progression free survival (mPFS); The secondary study endpoints are objective response rate (ORR), disease control rate (DCR), median overall survival time (mOS), and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1) The patient voluntarily participated in this study and signed an informed consent form; 2) Age>18 years old, both male and female; 3) Advanced stage unresectable or metastatic NSCLC (stage IIIB, IIIC, or IV) confirmed by histology or cytology, with the presence of EGFR 21 exon L858R mutation in the driving gene; 4) According to the criteria for evaluating the efficacy of solid tumors (RECIST 1.1), at least one measurable lesion is used as the target lesion; 5) The Eastern Cancer Collaborative Group's Physical State Score (ECOG PS) is 0 to 3 points; 6) Expected survival time is more than 3 months; 7) Newly treated patients who have not received systematic anti-tumor treatment in the past, including radiotherapy and chemotherapy, targeted and immunotherapy; 8) The main organ function meets the following standards within 7 days before treatment:(1) Blood routine examination standard (without blood transfusion within 14 days): ① Hemoglobin (HB) ≥ 90g/L; ② Absolute value of neutrophils (ANC) ≥ 1.5 × 109/L; ③ Platelet (PLT) ≥ 80 × 109/L.(2) Biochemical examination should meet the following standards: ① Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); ② Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5ULN, if accompanied by liver metastasis, ALT and AST ≤ 5ULN; ③ Serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance rate (CCr) ≥ 60ml/min.

Exclusion Criteria:

1. Mixed NSCLC containing other pathological components;
2. Poor blood pressure control (systolic blood pressure ≥ 150mmHg, diastolic blood pressure ≥ 100mmHg);
3. Imaging shows that the tumor invades important blood vessels, or the researcher determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies;
4. Have experienced arteriovenous thrombosis events within 6 months, such as cerebrovascular accidents, deep venous thrombosis, and pulmonary embolism in patients;
5. Patients with combined factors that affect oral medication, such as difficulty swallowing, gastrointestinal resection, chronic diarrhea, or intestinal obstruction;
6. Patients with symptomatic brain metastases;
7. Patients with severe and/or uncontrollable diseases, such as myocardial infarction, unstable angina, congestive heart failure, and severe uncontrollable arrhythmias within 6 months prior to enrollment;
8. Active or uncontrolled severe infections;
9. Severe liver dysfunction, cirrhosis, acute or chronic active hepatitis;
10. The urine routine results showed that the urine protein level was ≥++, and the 24-hour urine protein quantitative detection result was>1.0g;
11. Active pulmonary tuberculosis;
12. Pregnant or lactating women;
13. According to the judgement of the researchers, the subjects may have other factors that may cause the study to be terminated midway, such as other serious illnesses (including mental illness) requiring concurrent treatment, serious laboratory test abnormalities, and accompanying family and social factors, which may affect the safety of the subjects or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
median Progressive Free Survival (mPFS) | up to two years
  The time from the subject's initiation of treatment with anlotinib and aumolertinib to the occurrence of disease progression.

SECONDARY OUTCOMES:
objective response rate(ORR) | 6 to 8 weeks after the subjects used the investigational drugs
  The percentage of subjects who achieved complete remission or partial remission after 6 to 8 weeks of treatment with anlotinib and aumolertinib.
Disease control rate (DCR) | 6 to 8 weeks after the subjects used the investigational drugs
  The percentage of subjects whose tumors shrink or remain stable after 6 to 8 weeks of treatment with anlotinib and aumolertinib.
median Overall survival(mOS) | up to three years
  Median time from subjects' enrollment to death for any reasons. For subjects who are lost to follow-up before death, the last follow-up time will be calculated as the time of death.
Safety of combined therapy | up to two years
  Number of participants who had drug-related adverse reactions during the trial and the degree of adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Kunming University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheng Y, He Y, Li W, Zhang HL, Zhou Q, Wang B, Liu C, Walding A, Saggese M, Huang X, Fan M, Wang J, Ramalingam SS. Osimertinib Versus Comparator EGFR TKI as First-Line Treatment for EGFR-Mutated Advanced NSCLC: FLAURA China, A Randomized Study. Target Oncol. 2021 Mar;16(2):165-176. doi: 10.1007/s11523-021-00794-6. Epub 2021 Feb 5. PMID 33544337
- [Result] Lin B, Song X, Yang D, Bai D, Yao Y, Lu N. Anlotinib inhibits angiogenesis via suppressing the activation of VEGFR2, PDGFRbeta and FGFR1. Gene. 2018 May 15;654:77-86. doi: 10.1016/j.gene.2018.02.026. Epub 2018 Feb 14. PMID 29454091
- [Result] Xie C, Wan X, Quan H, Zheng M, Fu L, Li Y, Lou L. Preclinical characterization of anlotinib, a highly potent and selective vascular endothelial growth factor receptor-2 inhibitor. Cancer Sci. 2018 Apr;109(4):1207-1219. doi: 10.1111/cas.13536. Epub 2018 Mar 25. PMID 29446853
- [Result] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152
- [Result] Si X, Zhang L, Wang H, Zhang X, Wang M, Han B, Li K, Wang Q, Shi J, Wang Z, Cheng Y, He J, Shi Y, Chen W, Wang X, Luo Y, Nan K, Jin F, Li B, Chen Y, Zhou J, Wang D. Quality of life results from a randomized, double-blinded, placebo-controlled, multi-center phase III trial of anlotinib in patients with advanced non-small cell lung cancer. Lung Cancer. 2018 Aug;122:32-37. doi: 10.1016/j.lungcan.2018.05.013. Epub 2018 May 18. PMID 30032842
- [Result] Si X, Zhang L, Wang H, Zhang X, Wang M, Han B, Li K, Wang Q, Shi J, Wang Z, Cheng Y, Shi Y, Chen W, Wang X, Luo Y, Nan K, Jin F. Management of anlotinib-related adverse events in patients with advanced non-small cell lung cancer: Experiences in ALTER-0303. Thorac Cancer. 2019 Mar;10(3):551-556. doi: 10.1111/1759-7714.12977. Epub 2019 Jan 21. PMID 30666799
- [Result] Wang Z, Cheng Y, An T, Gao H, Wang K, Zhou Q, Hu Y, Song Y, Ding C, Peng F, Liang L, Hu Y, Huang C, Zhou C, Shi Y, Zhang L, Ye X, Zhang M, Chuai S, Zhu G, Hu J, Wu YL, Wang J. Detection of EGFR mutations in plasma circulating tumour DNA as a selection criterion for first-line gefitinib treatment in patients with advanced lung adenocarcinoma (BENEFIT): a phase 2, single-arm, multicentre clinical trial. Lancet Respir Med. 2018 Sep;6(9):681-690. doi: 10.1016/S2213-2600(18)30264-9. Epub 2018 Jul 17. PMID 30017884
- [Result] Zhou Q, Xu CR, Cheng Y, Liu YP, Chen GY, Cui JW, Yang N, Song Y, Li XL, Lu S, Zhou JY, Ma ZY, Yu SY, Huang C, Shu YQ, Wang Z, Yang JJ, Tu HY, Zhong WZ, Wu YL. Bevacizumab plus erlotinib in Chinese patients with untreated, EGFR-mutated, advanced NSCLC (ARTEMIS-CTONG1509): A multicenter phase 3 study. Cancer Cell. 2021 Sep 13;39(9):1279-1291.e3. doi: 10.1016/j.ccell.2021.07.005. Epub 2021 Aug 12. PMID 34388377